CLINICAL TRIAL: NCT07129720
Title: Assessment of a Molar-Incisor Hypomineralization Interventional Education Program on Knowledge, Attitude and Awareness Among a Group of Dental Interns.
Brief Title: Educational Program to Improve Dental Interns, Knowledge ,Attitude and Awareness Toward Molar Incisor Hypo-mineralization.
Acronym: MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, nada abd elmanem ahmed abo elsoud, BSC, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FU-MIH-EDU-2025-01
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Receiving Pre-Post Educational Intervention. (Experimental): Participants will receive a structured educational program on , MIH with pre- and post-intervention assessment.
  Interventions: Behavioral: Educational Program on MIH

INTERVENTIONS:
Behavioral: Educational Program on MIH — A 30-minute interactive educational session that includes a PowerPoint presentation, clinical images, and case-based discussions on Molar-Incisor Hypomineralization (MIH).
  The session covers the definition, eatiology , clinical features, diagnosis and evidence-based treatment options of MIH.
  The goal is to improve the participants' knowledge ,attitude and awareness . Evaluation will be conducted through pre- and post-intervention questionnaire.

SUMMARY:
This interventional, quasi experimental study aims to assess the effectiveness of an educational program on improving dental interns' knowledge, attitude and awareness regarding Molar-Incisor Hypo-mineralization (MIH).

A total of 200 dental interns from Future University will participate. A structured questionnaire will be administered before and after the educational intervention to measure changes in participants' knowledge , attitude and awareness.

The study seeks to evaluate whether targeted educational efforts can enhance clinical awareness and management approaches toward MIH among dental interns

DETAILED DESCRIPTION:
This study is designed as an interventional quasi experimental study . Educational research project conducted among dental interns at Future University.

The primary objective is to evaluate the impact of a structured educational program on the knowledge , awareness and attitude of dental interns regarding Molar-Incisor Hypo-mineralization (MIH).

A total of 200 dental interns will be invited to participate. The study will follow a pre-test/post-test design, in which participants will complete a validated questionnaire before and after attending the educational session.

The session will include a lecture covering the aetiology , clinical features, diagnosis, and management strategies of MIH.

Data collected will be analysed to determine if there are statistically significant improvements in knowledge ,attitude and awareness following the intervention. The results of this study may support the integration of targeted MIH education into undergraduate dental training to enhance future practitioners' ability to diagnose and manage MIH cases effectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be selected based on the following criteria.

A- Inclusion criteria:

* Dental interns currently enrolled at FUE in the study period.
* Assess to an internet-enabled device to complete the electronic questionnaire.
* Those who consented to participate in the study and completed the informed consent procedure.

B- Exclusion criteria:

* Dental students.
* Licensed Dentists.
* Incomplete or Duplicated Responses.
* Those who did not consent to participate.

Ages: 23 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
1ry Outcome To evaluate effectiveness of an educational program on knowledge, attitude and awareness regarding MIH among dental interns. | Baseline
  The survey consists of three sections to assess knowledge, attitude, and awareness toward Molar-Incisor Hypomineralization (MIH). The knowledge section includes 13 multiple-choice questions covering etiology, clinical features, diagnosis, and management of MIH. Each correct answer scores 1 point, with a total range of 0-13; higher scores indicate better knowledge. The attitude section contains 8 items rated on a 5-point Likert scale (Strongly Agree to Strongly Disagree), total range 8-40; higher scores indicate more positive attitudes. The awareness section includes 2 clinical case scenarios with structured questions; each correct answer scores 1 point, total range 0-2; higher scores reflect better awareness and diagnostic ability.

CONTACTS AND LOCATIONS:
Overall Officials: Abla A. Aly, Phd, Study Chair — Faculty of Dentistry, Future University in Egypt.; Eman A . Abdallah., Phd, Principal Investigator — Faculty of Dentistry, Future University in Egypt.
Locations (1):
- Faculty of Dentistry, Future University in Egypt, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The data collected during the study will be used solely for statistical analysis and reporting within the scope of this research project. No data will be made publicly available or shared with external researchers.